CLINICAL TRIAL: NCT01680848
Title: Assessment of Caries Diagnosis and Caries Treatment in Dental PBRN Japan
Status: Completed | Type: Observational
Sponsor: Dental PBRN Japan (Network)
Collaborators: Dental Practice-Based Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: E1157
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-08

CONDITIONS: Dental Caries
Keywords: Dental caries,; Caries diagnosis,; Caries treatment,; Caries risk,; Practice pattern,; Clinical epidemiology,; Dental Practice-Based Research Network
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to examine what methods Dental PBRN Japan dentists adopt for diagnosis, treatment, and prevention of dental caries.

DETAILED DESCRIPTION:
We conducted a cross-sectional study consisting of a questionnaire survey in Japan. We used the same questionnaire as used in the DPBRN Study, "Assessment of Caries Diagnosis and Caries Treatment".

ELIGIBILITY:
Inclusion Criteria:

* This study queried dentists working in outpatient dental practices who have affiliated with JDPBRN to investigate research questions and to share experiences and expertise (n = 282).

Exclusion Criteria:

* Dentist who doesn't perform some measure of restorative dentistry at their practice.

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are dentists who work in outpatient dental practices who have affiliated with Dental PBRN Japan
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Kakudate, DDS PhD MPH, Principal Investigator — Kyushu Dental University

IPD SHARING:
Plan to Share IPD: No
Currently, we have no plan.

REFERENCES:
- [Derived] Yokoyama Y, Kakudate N, Sumida F, Matsumoto Y, Gilbert GH, Gordan VV. Evidence-practice gap for dental sealant application: results from a dental practice-based research network in Japan. Int Dent J. 2016 Dec;66(6):330-336. doi: 10.1111/idj.12252. Epub 2016 Jul 28. PMID 27466073
- [Derived] Yokoyama Y, Kakudate N, Sumida F, Matsumoto Y, Gilbert GH, Gordan VV. Evidence-practice gap for in-office fluoride application in a dental practice-based research network. J Public Health Dent. 2016 Mar;76(2):91-7. doi: 10.1111/jphd.12114. Epub 2015 Jul 31. PMID 26235360
- [Derived] Kakudate N, Sumida F, Matsumoto Y, Yokoyama Y, Riley JL 3rd, Gilbert GH, Gordan VV. Dentists' decisions to conduct caries risk assessment in a Dental Practice-Based Research Network. Community Dent Oral Epidemiol. 2015 Apr;43(2):128-34. doi: 10.1111/cdoe.12127. Epub 2014 Sep 1. PMID 25175077
- [Derived] Kakudate N, Sumida F, Matsumoto Y, Yokoyama Y, Gilbert GH, Gordan VV. Patient age and dentists' decisions about occlusal caries treatment thresholds. Oper Dent. 2014 Sep-Oct;39(5):473-80. doi: 10.2341/13-141-C. Epub 2014 May 8. PMID 24809540
- [Derived] Yokoyama Y, Kakudate N, Sumida F, Matsumoto Y, Gilbert GH, Gordan VV. Dentists' dietary perception and practice patterns in a dental practice-based research network. PLoS One. 2013;8(3):e59615. doi: 10.1371/journal.pone.0059615. Epub 2013 Mar 25. PMID 23536883
- [Derived] Kakudate N, Sumida F, Matsumoto Y, Manabe K, Yokoyama Y, Gilbert GH, Gordan VV. Restorative treatment thresholds for proximal caries in dental PBRN. J Dent Res. 2012 Dec;91(12):1202-8. doi: 10.1177/0022034512464778. Epub 2012 Oct 9. PMID 23053847

RESULTS

PARTICIPANT FLOW:
Groups:
- JDPBRN Dentists: Dentists working in outpatient dental practice (n=282) who were affiliated with the JDPBRN and who indicated that they do at least some restorative dentistry.
Period: Overall Study
Arm/Group | JDPBRN Dentists
Started | 282
Completed | 189
Not Completed | 93

BASELINE CHARACTERISTICS:
Groups:
- JDPBRN Dentists: Dentists working in outpatient dental practice (n=282) who were affiliated with the JDPBRN and who indicated that they do at least some restorative dentistry.
  The JDPBRN aims to allow dentists to investigate research questions and share experiences and expertise and recruited its members from the JDPBRN website.
Arm/Group | JDPBRN Dentists
Number analyzed (Participants) | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 189
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 186
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Participants were recruited from the JDPBRN Web site and mailings if they indicated that they perform some measure of restorative dentistry at their practice.
  participants
    Japan | 189
The mean number of years elapsed since graduation from dental school [Mean (Standard Deviation); unit: years] | 18.5 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Indicate Surgical Intervention
Time Frame: Up to 24 months
Measure: Number; unit: percentage of the dentists
Groups:
- High Caries Risk: The proportion of dentists who indicated surgical intervention into enamel was 74% (N = 138) in the high-caries-risk scenario.
Arm/Group | High Caries Risk
Number analyzed (Participants) | 187
percentage of the dentists | 74

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed.
Groups:
- This is an Observational Study: This is an observational study. We don't have two arms.
Arm/Group | This is an Observational Study
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No